CLINICAL TRIAL: NCT07339852
Title: Implementation and Evaluation of a Pharmacist-led Diabetes Care Pathway in Alberta Community Pharmacies.
Acronym: D-PATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00145395
Record Dates: First submitted 2025-06-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidaemia
Keywords: diabetes; pharmacist; pathway; shared decision making
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led care pathway (Experimental): Participants in the intervention arm will receive the care using a shared decision-making pharmacist care pathway approach designed to guide type 2 diabetes management to achieve target A1C levels and reduce the risk of diabetes-related complications. The pharmacist care pathway is modelled after the Canadian Diabetes Association Guidelines. This pathway (tool) will be built into a computer web-based program and include step-by-step, algorithm-guided patient assessment to achieve target A1C levels and reduce the risk of diabetes-related complications. This will occur through follow-ups every 6 weeks for six months duration.
  Interventions: Other: Pharmacist-led diabetes care pathway
- Usual Care (No Intervention): The control group will involve facilitated relay of information to participants' family physician or nurse practitioner. Participants in the control group will have their pharmacist collect information informing the patient's current diabetes control. Participants will then be given a letter that contains their A1C value, and they will be advised to present it to their family physician or nurse practitioner. No specific suggestions for diabetes management will be detailed in the letter. In the case where the patient does not have a family physician or nurse practitioner, they will be referred to a physician walk-in clinic. A follow-up appointment will be booked for all participants in the control group at 3-months to discuss dietary and lifestyle interventions in the management of type 2 diabetes to maintain participant interest in the study and again at 6-months' time for a final visit.

INTERVENTIONS:
Other: Pharmacist-led diabetes care pathway — articipants in the intervention arm will receive the care using a shared decision-making pharmacist care pathway approach designed to guide type 2 diabetes management to achieve target A1C levels and reduce the risk of diabetes-related complications. The pharmacist care pathway is modelled after the Canadian Diabetes Association Guidelines22. This pathway (tool) will be built into a computer web-based program and include step-by-step, algorithm-guided patient assessment to achieve target A1C levels and reduce the risk of diabetes-related complications. This will occur through follow-ups every 6 weeks for six months duration.
  Arms: Pharmacist-led care pathway

SUMMARY:
As of 2024, nine percent of Albertans are living with Type 2 diabetes, which increases their risk for cardiovascular disease, stroke, blindness, and kidney failure. Unfortunately, less than half of patients have controlled Type 2 diabetes. We are well aware of the factors which lead to worsening diabetes, but need to give people more support to help them manage their diabetes. Pharmacists are respected health care professionals who are often easier to see that doctors and can help people with diabetes to stay as healthy as possible.

This research project aims to see whether a pharmacist service can help improve diabetes management in people with type 2 diabetes compared to usual care from their family physician or nurse practitionner. The potential impact of this project is to empower people with type 2 diabetes to understand their condition, it's management, and to achieve target blood sugar levels, which will ultimately reduce the risk of diabetes-related complications.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 years or older.
2. Individuals with type 2 diabetes.
3. Individuals with type 2 diabetes not reaching HbA1c target of under 7.0%

Exclusion Criteria:

1. Individuals with type 1 diabetes, gestational diabetes, or other forms of diabetes that are not type 2 diabetes.
2. Pregnant individuals.
3. Individuals at their HbA1c target (HbA1c under 7.0%) or those with a limited life expectancy, frailty, or lack hypoglycemic awareness (i.e., those with an A1c target above 7.0%) .
4. Individuals unable to provide consent or who are unwilling to attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
A1C change | Up to 6 months
  The primary outcome is the difference in change in A1C calculated from baseline to the end of the study (up to six months) between the intervention and control groups.

SECONDARY OUTCOMES:
Estimated cardiovascular risk | Up to 6 months.
  The primary outcome is the difference in change in estimated CV risk from baseline to the end of the study (up to six months) between the intervention and control groups.
Blood Pressure | Up to 6 months.
  The difference in change in blood pressure from baseline to the end of the study (up to six months) between the intervention and control groups.
LDL cholesterol concentration | Up to 6 months.
  The difference in change in serum LDL-cholesterol concentration from baseline to the end of the study (up to six months) between the intervention and control groups
Influenza vaccination | Up to 6 months.
  The difference in the proportion of participants who receive their influenza vaccination from baseline to the end of the study (up to six months) between the intervention and control groups.
Pneumococcal vaccination | Up to 6 months
  The difference in the proportion of participants who receive their pneumococcal vaccination from baseline to the end of the study (up to six months) between the intervention and control groups.
Foot exam | Up to 6 months
  The difference in the proportion of participants who complete foot exams from baseline to the end of the study (up to six months) between the intervention and control groups.
Eye Exam | Up to 6 months.
  The difference in the proportion of participants who complete eye exams from baseline to the end of the study (up to six months) between the intervention and control groups.
Renal function screening | Up to 6 months.
  The difference in the proportion of participants who complete renal function screening (glomerular filtraion rate, albumin to creatinine ratio) from baseline to the end of the study (up to six months) between the intervention and control groups.
Vascular Protection | Up to 6 months.
  The difference in the proportion of participants who have guideline-based vascular protection in place from baseline to the end of the study (up to six months) between the intervention and control groups.
Pharmacist prescribed prescription medications | Up to 6 months.
  Pharmacist prescribing or changing the dose of medications from baseline to the end of the study (up to six months) between the intervention and control groups.
Pharmacist provided education on lifestyle factors | Up to 6 months
  Education on lifestyle factors (tobacco cessation, diet, exercise) from baseline to the end of the study (up to six months) between the intervention and control groups.
Pharmacist provided education on medications and importance of adherence. | Up to 6 months
  Pharmacist intervention of providing education on medications and importance of adherence from baseline to the end of the study (up to six months) between the intervention and control groups.
Laboratory Monitoring | Up to 6 months.
  The difference in the proportion of participants who attend the laboratory for routine monitoring from baseline to the end of the study (up to six months) between the intervention and control groups.
Continuous Glucose Monitoring | Up to 6 months.
  The difference in the proportion of participants who use continuous glucose monitoring devices from baseline to the end of the study (up to six months) between the intervention and control groups.
Yield of enrolment approaches | Up to 6 months.
  The yield from each enrolment approach used (active case-finding approach vs. passive approaches such as when the patient attends the pharmacy to collect a prescription medication or through patient self-identification).
Yield of enrollment by pharmacy type | Up to 6 months.
  Yield of enrollment by clinic or non-clinic pharmacy type.
Shared-decision making uptake | Up to 6 months.
  Extent to which shared decision making was achieved in the intervention as measured by the validated Shared Decision Making 9-item Questionnaire (SDM-Q-9) tool. The minimum score is 0 and the maximum score is 45, where a higher score indicates a greater subjective level of shared decision making.
Patient satisfaction - standard | Up to 6 months.
  Patient satisfaction as measured by the diabetes treatment satisfaction questionnaire standard (DTSQs). The standard version of the DTSQ consists of eight questions on a 0-6 Likert scale (where 0 is very dissatisfied and 6 is very satisfied). Minimum score = 0, maximum score = 48.
Patient satisfaction - change | Up to 6 months.
  Patient satisfaction as measured by the diabetes treatment satisfaction questionnaire change (DTSQc). It is designed to overcome ceiling effects, where satisfaction is already high, by allowing for more precise reporting of improvements or declines, and thus must be used alongside the DTSQs to understand both the absolute satisfaction level and the change over time.
  The change version of the DTSQ consists of eight questions on a 0-6 Likert scale (where 0 is very dissatisfied and 6 is very satisfied). Minimum score = 0, maximum score = 48.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, BScPharm, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT07339852/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT07339852/ICF_001.pdf